CLINICAL TRIAL: NCT02259543
Title: Conditioning of Root Surfaces With Citric Acid and Tetracycline for Different Application Times Improves the Outcomes of Root Coverage by Subepithelial Connective Tissue Graft: a Randomized Clinical Trial.
Brief Title: Root Biomodification With Citric Acid and Tetracycline Improves the Outcomes of Root Coverage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Adriana Campos Passanezi SantAna, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 018/2010
Record Dates: First submitted 2014-09-28; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Gingival Recession
Keywords: gingival recession; soft tissue; root biomodification; root coverage; citric acid; tetracycline
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- G0 (No Intervention): Root decontamination performed by scaling and root planing followed by rinsing with saline solution during the treatment of recession defects by subepithelial connective tissue graft (SCTG). Control group.
- G90 (Active Comparator): Root conditioning with citric acid+tetracycline solution (1:1) for 90 seconds after scaling and root planing, followed by rinsing with saline solution for root decontamination during the treatment of recession defects by subepithelial connective tissue graft (SCTG).
  Interventions: Other: Root conditioning with citric acid+tetracycline solution
- G180 (Active Comparator): Root conditioning with citric acid+tetracycline solution (1:1) for 180 seconds after scaling and root planing, followed by rinsing with saline solution for root decontamination during the treatment of recession defects by subepithelial connective tissue graft (SCTG).
  Interventions: Other: Root conditioning with citric acid+tetracycline solution

INTERVENTIONS:
Other: Root conditioning with citric acid+tetracycline solution — Application of a citric acid + tetracycline gel solution (1:1) for decontamination of root surfaces during the treatment of recession defects by subepithelial connective tissue graft
  Arms: G180; G90

SUMMARY:
The aim of this study is to investigate the effects of the application of a citric acid + tetracycline gel solution during 90 or 180 seconds compared to no conditioning in the outcomes of treatment of Miller's class I or II recession defects by subepithelial connective tissue graft.

DETAILED DESCRIPTION:
Adult patients showing Miller's class I or II recession defects requiring root coverage were recruited to participate in the study. All patients were submitted to non surgical periodontal therapy consisting of scaling and root planing, prophylaxis, and oral hygiene instruction in order to reduce/eliminate gingival inflammation. After that, patients were randomly allocated to three different treatment groups based on root conditioning: G0- no conditioning; G90- root conditioning for 90 seconds; G180- root conditioning for 180 seconds. Allocation was defined by a software. Root coverage was performed by subepithelial connective tissue graft (SCTG) in all treated sites by the same operator, who performed the indicated root treatment. Periodontal parameters were investigated at baseline and at 1, 3, 6 and 12 months post-operatively by a blinded trained expertise different from operator and included: pocket depth, recession height, clinical attachment level, width of keratinized gingiva, sulcular bleeding index and plaque index. Hypersensitivity at recession sites was also investigated at baseline and at 7 days, 14 days, 1, 3, 6 and 12 months after treatment according to visual analogic scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* presence of Miller's class I or II recession extending 2-5 mm apical to CEJ requiring root coverage for the following reasons: esthetics, progression of recession or hypersensitivity.

Exclusion Criteria:

* smokers;
* pregnants;
* routine use of anti-convulsants, anti-hypertensive or cyclosporine;
* uncontrolled systemic diseases (e.g.: diabetes mellitus);
* systemic conditions that requires antibiotic prophylaxis (e.g.: history of bacterial endocarditis; rheumatoid arthritis; prosthetic valves);
* antibiotics, steroidal or non-steroidal anti-inflammatory intake in the 6-month previous period.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
percentage of root coverage (%REC) | one year
  Percentage of root coverage obtained at 1 year after procedure. Represented by the difference of baseline recession height and final recession height divided by baseline recession height multiplied by 100 (in percentage).

SECONDARY OUTCOMES:
reduction in recession height | one year
  Linear difference between final recession height and baseline recession height, measured by a millimeter periodontal probe as the distance from cementum-enamel junction and gingival margin at the center of recession defect (in mm).
increase in the width of keratinized gingiva | one year
  Linear difference between final and baseline width of keratinized gingiva. Measured with a millimeter periodontal problem as the distance from gingival margin to mucogingival junction (in mm).
gain in clinical attachment level | one year
  Linear difference between final and baseline clinical attachment level. Measured with a millimeter periodontal probe as the distance from cementum-enamel junction and the bottom of the sulcus or pocket (in mm).

OTHER OUTCOMES:
reduction in probing depth | one year
  Linear difference of final and baseline probing pocket measurements. Measured with a millimeter periodontal probe as the distance between gingival margin and the bottom of the sulcus or pocket (in mm).
reduction in bleeding index | one year
  Difference in the presence (score 1) or absence (0) of bleeding on probing, up to 10 seconds after removal of the probe from the sulcus (index; percentage)
reduction in plaque index | one year
  Difference in the presence (score 1) or absence (score 0) of plaque accumulation, visually determined (index; percentage)

CONTACTS AND LOCATIONS:
Overall Officials: João Paulo C Barros, Master, Principal Investigator — Graduation student
Locations (1):
- School of Dentistry at Bauru- University of São Paulo; Clinics of Periodontics, Bauru, São Paulo, Brazil